CLINICAL TRIAL: NCT03268616
Title: Investigation of the Correlation of Surface Respiratory EMG With Esophageal Diaphragm EMG
Brief Title: Analyse the Correlation Between sEMG and EMGdi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Lin Lin, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 487201278
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: COPD
Keywords: neural respiratory drive; noninvasive positive pressure ventilation; electromyography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Subjects (Experimental): increase the inspiratory threshold load step by step(30%-80%MIP),in order to increase neural respiratory drive.
  Interventions: Device: inspiratory threshold load device and NPPV
- Sever COPD Patients (Experimental): increase the pressure support ventilation step by step, in order to decrease neural respiratory drive.
  Interventions: Device: inspiratory threshold load device and NPPV

INTERVENTIONS:
Device: inspiratory threshold load device and NPPV — before experiment ,every subject use a flanged mouthpiece attached to a manually operated occlusion valve in order to measure maximal inspiratory pressure (MIP)at functional residual capacity .
  healthy subjects:increase the pressure in a water-sealed inspiratory threshold loading device in order to increase the neural respiratory drive.
  COPD patients:increase the pressure in a non-invasive positive pressure ventilation in order to decrease the neural respiratory drive

SUMMARY:
The most significant pathophysiology change of COPD patients is persistent incompletely reversible airflow obstruction and increased lung volume. As a result, the work of breathing(WB) and neural respiratory drive (NRD)increased. Noninvasive positive pressure ventilation (NPPV) can reduce the load of respiratory muscles. Detection of NRD can be the index of monitoring for titration of optimal level of ventilator support in the future. As electromyography(EMG) is the most reliable measurement in evaluating NRD that can be used for human. Currently the standard method for evaluation of NRD with EMG is using esophageal multi-paired electrodes catheter(EMGdi) ,it is reliable but invasive .Surface respiratory EMG (sEMG）is a noninvasive measurement. Although it subjected to contamination and less sensitive, recently, advance in technology with multiple pair of surface electrodes is possible to sufficient signals for evaluation of NRD.So the investigator compare the NRD measured by EMGdi and sEMG,and consider that the correlation between them is well in different levels.

DETAILED DESCRIPTION:
The most significant pathophysiology change of COPD patients is persistent incompletely reversible airflow obstruction and increased lung volume. As a result, the work of breathing (WB) and neural respiratory drive (NRD) increased. Noninvasive positive pressure ventilation (NPPV) is the first-line treatment in acute exacerbation of COPD (AECOPD). One of the mechanisms is to reduce the load of respiratory muscles. It has been reported that NRD decreased in response to increase of pressure support. Detection of NRD can be the index of monitoring for titration of optimal level of ventilator support in the future.

NRD can be measured with minute ventilation, inspiratory pressure change、mean inspiration flow and electromyography(EMG) of inspiratory muscles. However, the first three methods are subjected to the influenced of lung volume, airway resistance and compliance of respiratory system. So, electromyography is the most reliable measurement in evaluating NRD that can be used for human. Currently the standard method for evaluation of NRD with EMG is using esophageal multi-paired electrodes catheter ,since it is far away from chest wall and close to diaphragm , so the contamination from other respiratory muscles can be reduced .However, catheter placement into esophagus is necessary for this measurement, which limits its use in daily practice. Surface respiratory EMG is a noninvasive measurement. Although it subjected to contamination and less sensitive, recent advance in technology with multiple pair of surface electrodes, including surface diaphragm EMG、parasternal EMG and so on, it is possible to sufficient signals for evaluation of NRD. It has been the hot topics of research recently due to its noninvasive, easiness of use and appropriate for continuing monitor.

Purpose：

1. To explore the feasibility of surface respiratory electromyography and its correlation with esophageal EMG in conditions of different level of respiratory central drive.
2. To investigate the dynamic change esophageal EMG and surface EMG in response to increase of pressure support level during noninvasive ventilation, in order to evaluate the feasibility of using surface EMG for titration of pressure support during noninvasive ventilation.

Methodology:

1. Electromyography: Multi-paired electrodes esophageal catheter was used for detection of esophageal diaphragm electromyography (EMGdi); Surface electrodes for left and right diaphragm and parasternal muscle were used to detect surface electromyography (sEMG).
2. Monitoring of respiratory physiology parameters: Pneumotachometer and differential pressure transducer were used for measurement of respiratory flow and pressures. lung volume change was calculated with integration of flow.
3. Regulate neural respiratory drive:1.in normal volunteer,increase the inspiratory threshold load step by step(30%-80%MIP),in order to increase neural respiratory drive;2.in sever COPD patients,increase the pressure support ventilation step by step, in order to decrease neural respiratory drive.
4. Methods for adjustment of respiratory central drive: (1) The increase of respiratory central drive was induced by inspiratory threshold load step by step (30%-80%MIP) in normal volunteer. (2) The reduction of respiratory central drive was induced by stepwise increase of pressure support level with noninvasive ventilation in COPD patients.

Analysis and statistics:

1. The correlation between sEMG and EMGdi at different level of respiratory central drive was analyzed with Pearson correlation analysis. The change of Ventilation central drive coupling was calculated.
2. In COPD patients, the change of respiratory central drive in response to increase of pressure support level (IPAP increase from 8cmH2O to 20cmH2O) during NPPV was evaluated.
3. The feasibility using sEMG as guidance for adjustment of pressure support level during NPPV was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* normal cardio-pulmonary function
* without low inspiratory muscle strength
* non-smoker
* without history of the nervous system and respiratory system disease
* sever to very severe stable stage

Exclusion Criteria:

* systemic application of corticosteroids nearly 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-07-02 (Actual)

PRIMARY OUTCOMES:
correlation between sEMG and EMGdi | through study completion, an average of 5 hours
  the correlation between sEMG and EMGdi at different level of respiratory central drive was analyzed with Pearson correlation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitelaw WA, Derenne JP. Airway occlusion pressure. J Appl Physiol (1985). 1993 Apr;74(4):1475-83. doi: 10.1152/jappl.1993.74.4.1475. PMID 8514660
- [Background] Luo YM, Moxham J, Polkey MI. Diaphragm electromyography using an oesophageal catheter: current concepts. Clin Sci (Lond). 2008 Oct;115(8):233-44. doi: 10.1042/CS20070348. PMID 18782085
- [Background] Reilly CC, Ward K, Jolley CJ, Lunt AC, Steier J, Elston C, Polkey MI, Rafferty GF, Moxham J. Neural respiratory drive, pulmonary mechanics and breathlessness in patients with cystic fibrosis. Thorax. 2011 Mar;66(3):240-6. doi: 10.1136/thx.2010.142646. Epub 2011 Feb 1. PMID 21285244
- [Background] Laghi F, Shaikh HS, Morales D, Sinderby C, Jubran A, Tobin MJ. Diaphragmatic neuromechanical coupling and mechanisms of hypercapnia during inspiratory loading. Respir Physiol Neurobiol. 2014 Jul 1;198:32-41. doi: 10.1016/j.resp.2014.03.004. Epub 2014 Apr 16. PMID 24747754
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Wanke T, Lahrmann H, Formanek D, Zwick H. Effect of posture on inspiratory muscle electromyogram response to hypercapnia. Eur J Appl Physiol Occup Physiol. 1992;64(3):266-71. doi: 10.1007/BF00626290. PMID 1563372
- [Result] Jolley CJ, Luo YM, Steier J, Reilly C, Seymour J, Lunt A, Ward K, Rafferty GF, Polkey MI, Moxham J. Neural respiratory drive in healthy subjects and in COPD. Eur Respir J. 2009 Feb;33(2):289-97. doi: 10.1183/09031936.00093408. Epub 2008 Oct 1. PMID 18829678
- [Result] Li Y, Li YH, Li S, Luo YW, Xiao R, Huang YX, Huang JL, Chen YT, Zhi RC, Chen X. Efficiency of neural respiratory drive for the assessment of bronchodilator responsiveness in patients with chronic obstructive pulmonary disease: an exploratory study. J Thorac Dis. 2016 May;8(5):958-65. doi: 10.21037/jtd.2016.03.70. PMID 27162672
- [Result] Murphy PB, Kumar A, Reilly C, Jolley C, Walterspacher S, Fedele F, Hopkinson NS, Man WD, Polkey MI, Moxham J, Hart N. Neural respiratory drive as a physiological biomarker to monitor change during acute exacerbations of COPD. Thorax. 2011 Jul;66(7):602-8. doi: 10.1136/thx.2010.151332. Epub 2011 May 19. PMID 21597112
- [Result] Suh ES, Mandal S, Harding R, Ramsay M, Kamalanathan M, Henderson K, O'Kane K, Douiri A, Hopkinson NS, Polkey MI, Rafferty G, Murphy PB, Moxham J, Hart N. Neural respiratory drive predicts clinical deterioration and safe discharge in exacerbations of COPD. Thorax. 2015 Dec;70(12):1123-30. doi: 10.1136/thoraxjnl-2015-207188. Epub 2015 Jul 20. PMID 26194996
- [Result] Jensen D, O'Donnell DE, Li R, Luo YM. Effects of dead space loading on neuro-muscular and neuro-ventilatory coupling of the respiratory system during exercise in healthy adults: implications for dyspnea and exercise tolerance. Respir Physiol Neurobiol. 2011 Dec 15;179(2-3):219-26. doi: 10.1016/j.resp.2011.08.009. Epub 2011 Aug 22. PMID 21888993
- [Result] Duiverman ML, van Eykern LA, Vennik PW, Koeter GH, Maarsingh EJ, Wijkstra PJ. Reproducibility and responsiveness of a noninvasive EMG technique of the respiratory muscles in COPD patients and in healthy subjects. J Appl Physiol (1985). 2004 May;96(5):1723-9. doi: 10.1152/japplphysiol.00914.2003. Epub 2003 Dec 5. PMID 14660508
- [Result] Maarsingh EJ, van Eykern LA, Sprikkelman AB, Hoekstra MO, van Aalderen WM. Respiratory muscle activity measured with a noninvasive EMG technique: technical aspects and reproducibility. J Appl Physiol (1985). 2000 Jun;88(6):1955-61. doi: 10.1152/jappl.2000.88.6.1955. PMID 10846005
- [Result] Nava S, Ambrosino N, Rubini F, Fracchia C, Rampulla C, Torri G, Calderini E. Effect of nasal pressure support ventilation and external PEEP on diaphragmatic activity in patients with severe stable COPD. Chest. 1993 Jan;103(1):143-50. doi: 10.1378/chest.103.1.143. PMID 8417869
- [Result] Reilly CC, Jolley CJ, Ward K, MacBean V, Moxham J, Rafferty GF. Neural respiratory drive measured during inspiratory threshold loading and acute hypercapnia in healthy individuals. Exp Physiol. 2013 Jul;98(7):1190-8. doi: 10.1113/expphysiol.2012.071415. Epub 2013 Mar 15. PMID 23504646
- [Result] Ju C, Chen R. Factors associated with impairment of quadriceps muscle function in Chinese patients with chronic obstructive pulmonary disease. PLoS One. 2014 Feb 18;9(2):e84167. doi: 10.1371/journal.pone.0084167. eCollection 2014. PMID 24558357
- [Result] De Troyer A. Inspiratory elevation of the ribs in the dog: primary role of the parasternals. J Appl Physiol (1985). 1991 Apr;70(4):1447-55. doi: 10.1152/jappl.1991.70.4.1447. PMID 1958250
- [Result] Cardoso DM, Fregonezi GA, Jost RT, Gass R, Alberton CL, Albuquerque IM, Paiva DN, Barreto SS. Acute effects of Expiratory Positive Airway Pressure (EPAP) on different levels in ventilation and electrical activity of sternocleidomastoid and parasternal muscles in Chronic Obstructive Pulmonary Disease (COPD) patients: a randomized controlled trial. Braz J Phys Ther. 2016 Nov-Dec;20(6):525-534. doi: 10.1590/bjpt-rbf.2014.0190. Epub 2016 Sep 16. PMID 27683840
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Result] Thys F, Roeseler J, Reynaert M, Liistro G, Rodenstein DO. Noninvasive ventilation for acute respiratory failure: a prospective randomised placebo-controlled trial. Eur Respir J. 2002 Sep;20(3):545-55. doi: 10.1183/09031936.02.00287402. PMID 12358327
- [Result] Kohnlein T, Windisch W, Kohler D, Drabik A, Geiseler J, Hartl S, Karg O, Laier-Groeneveld G, Nava S, Schonhofer B, Schucher B, Wegscheider K, Criee CP, Welte T. Non-invasive positive pressure ventilation for the treatment of severe stable chronic obstructive pulmonary disease: a prospective, multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2014 Sep;2(9):698-705. doi: 10.1016/S2213-2600(14)70153-5. Epub 2014 Jul 24. PMID 25066329
- [Result] Casanova C, Celli BR, Tost L, Soriano E, Abreu J, Velasco V, Santolaria F. Long-term controlled trial of nocturnal nasal positive pressure ventilation in patients with severe COPD. Chest. 2000 Dec;118(6):1582-90. doi: 10.1378/chest.118.6.1582. PMID 11115443
- [Result] Dreher M, Storre JH, Schmoor C, Windisch W. High-intensity versus low-intensity non-invasive ventilation in patients with stable hypercapnic COPD: a randomised crossover trial. Thorax. 2010 Apr;65(4):303-8. doi: 10.1136/thx.2009.124263. PMID 20388753
- [Result] Zhang J, Luo Q, Zhang H, Chen R. Effect of noninvasive proportional assist vs pressure support ventilation on neuroventilatory coupling in chronic obstructive pulmonary patients with hypercapnia. Intensive Care Med. 2014 Sep;40(9):1390-1. doi: 10.1007/s00134-014-3378-5. Epub 2014 Jun 27. No abstract available. PMID 24968715
- [Result] Passam F, Hoing S, Prinianakis G, Siafakas N, Milic-Emili J, Georgopoulos D. Effect of different levels of pressure support and proportional assist ventilation on breathing pattern, work of breathing and gas exchange in mechanically ventilated hypercapnic COPD patients with acute respiratory failure. Respiration. 2003 Jul-Aug;70(4):355-61. doi: 10.1159/000072897. PMID 14512669